CLINICAL TRIAL: NCT06821620
Title: Interaction of MTNR1B Genotype and Type of Breakfast (Protein-enriched v Carbohydrate-rich) on Postprandial Glucose Response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SMU_ETHICS_2023-24_626
Record Dates: First submitted 2024-08-01; First posted 2025-02-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Breakfast

STUDY DESIGN:
Who Masked: Participant
Masking Description: Breakfast condition - high carbohydrate or protein enriched
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein enriched breakfast (Experimental)
  Interventions: Dietary Supplement: Breakfast
- High carbohydrate breakfast (Active Comparator)
  Interventions: Dietary Supplement: Breakfast

INTERVENTIONS:
Dietary Supplement: Breakfast — Breakfast in one condition will be high carbohydrate and in the other protein enriched

SUMMARY:
The risk version of the MTNR1B gene (which codes for a melatonin receptor) has been associated with type II diabetes (T2D) and associated physiological markers. People with the risk version of the gene have reduced secretion of insulin when melatonin levels are high (between evening and morning) and impaired glucose tolerance when they eat late. Previous research suggests eating a protein enriched breakfast can improve glucose response. Therefore, the present study will investigate if the version of the MTNR1B gene that people have is associated with their glucose response after breakfast. Also, whether a protein enriched breakfast improves glucose response in participants with the risk version of the gene. Measures of glucose response collected over the two-week duration of the study will be compared between groups with the different versions of the gene. These findings can be used to provide personalised nutrition advice which may reduce the risk of T2D.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-48 years*, not diabetic, not sleep disorder, not relevant medication (weight loss, sleeping, melatonin), not restricted diet, not allergic to oats, milk, wheat, barley or soya, not implanted medical device, such as pacemakers.

Exclusion Criteria:

* aged < 18 or > 48 years, diabetic, sleep disorder, eating disorder, taking relevant medication (weight loss, sleeping, melatonin), following a restricted diet, implanted medical device, such as pacemakers.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Glucose response | 120 minutes
  Area under the curve

SECONDARY OUTCOMES:
CGM metrics - mean glucose | 14 days
  mean glucose for 14 days measured using (FreeStyle Libre Pro iQ Continuous Glucose Monitoring System)
CGM metrics - Time in range | 14 days
  Time in range for 14 day period (FreeStyle Libre Pro iQ Continuous Glucose Monitoring System)
CGM metrics - glycaemic variability | 14 days
  glycaemic variability for 14 day period (FreeStyle Libre Pro iQ Continuous Glucose Monitoring System)

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No